CLINICAL TRIAL: NCT02608593
Title: Breast Reconstruction Outcomes With and Without StratticE (BROWSE)
Brief Title: Breast Reconstruction Outcomes With and Without StratticE
Acronym: BROWSE
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: LifeCell (Industry)
Responsible Party: Sponsor
Other Study IDs: BROWSE
Record Dates: First submitted 2015-10-26; First posted 2015-11-18 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — strattice

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Implant reconstruction with Strattice: Women having immediate breast reconstruction with partial or total Strattice cover
  Interventions: Procedure: Strattice
- Implant reconstruction without Strattice: Women having immediate implant based breast reconstruction where no Strattice has been used

INTERVENTIONS:
Procedure: Strattice — Implant based reconstruction with strattice cover of part or all of implant
  Groups: Implant reconstruction with Strattice

SUMMARY:
Approximately 4,000 women undergo a mastectomy for breast cancer each year in the UK and around 1,500 will have an immediate breast reconstruction. Approximately half of these ladies will have an implant-based breast reconstruction, of which many have an "implant-assisted" breast reconstruction with an Acellular Dermal Matrix.

Strattice™ is an Acellular Dermal Matrix (a pig skin product) made by Acelity. It is used to cover and disguise the lower part of the breast implant. Acellular Dermal Matrices have only been widely used for the last eight years and long-term outcomes for women who have had this form of reconstruction are lacking. Despite this, it is one of the most commonly offered methods of breast reconstruction in the UK for both ladies with a diagnosis of breast cancer and in the risk-reduction setting.

The objective of this study is to assess long-term outcomes of Strattice™-based breast reconstructions in multiple Breast Surgery Centres across the UK. This will be a case-control study comparing women who have had an immediate implant-based breast reconstruction with Strattice™ (case) or without (control). This will be achieved by review and analysis of retrospective data from patients who have undergone immediate breast reconstruction using implants with or without Strattice™ following either a diagnosis breast cancer or for risk-reduction. In addition there will be a prospective clinical assessment of the reconstruction outcomes. Outcomes assessed will include complications, surgical re-interventions and aesthetic results. These will be related to co-morbid conditions and other risk factors. Data will also be collected on unplanned interventions associated with a cost, if available.

DETAILED DESCRIPTION:
Primary Outcome The primary outcome measure will be unexpected loss of the implant.

Secondary Outcomes

To investigate short and long-term outcomes with Strattice™ including:

* Quality of Life
* In-patient treatment costs
* Ipsilateral Revision rates
* Aesthetic outcome
* Breast reconstruction softness (Tonometry)
* Regional pain
* Loco-regional recurrence
* Effect of radiotherapy
* Complications - (seroma drainage, skin necrosis/ wound breakdown)

Study Design

* All patients who have had an immediate implant-based breast reconstruction will be identified from prospective databases.
* Patients will be invited to enter the research study by post. The invitation letter will include: an offer to take part in the study, a Patient Information Leaflet, a Stamped addressed envelope and an Accept/Decline outcome form.
* If they fail to respond, patients will be re-contacted on one further occasion, in the same manner, after approximately two months.
* Patients will be invited to attend a clinical appointment at the Breast Surgery Centre where their reconstruction was performed. Here they will see a clinical researcher in the presence of a clinic nurse and consent to participate in the study.
* Patients will be asked to undergo a clinical assessment, Tonometry (measurement of breast reconstruction softness) and medical photography. The data obtained from this will be anonymised and inputted into a database for analysis.
* Patients will receive a postal questionnaire following the clinic visit asking them about the "Patient Reported Outcomes" of their reconstruction. (This will not be performed at the clinic visit in an attempt to avoid bias). They will receive a further follow-up questionnaire 12 months later.
* The medical records of patients will be reviewed to assess outcomes including complications from surgery.
* If a patient does not consent for the prospective part of the study, a retrospective audit of their notes for implant loss, revisions and complications will be performed
* All data will be collected on Case Report Forms. Study numbers will be allocated, and linked-anonymised data inputted into a database on a NHS computer for analysis.
* Medical records, including clinic letters, nursing records and anaesthetic charts will be reviewed to collect data on:

  * Patient demographics (age, BMI, comorbidities and smoking history at time of surgery)
  * Surgical details (operation type, operation time, mastectomy weight, implant size/type)
  * Details on cancer outcome and adjuvant therapies
  * Post-operative complications (including need for reoperation, prolonged healing, loss of implant)
* Additional prospective data analysed will include:

  * Patient Reported Outcome questionnaire results
  * Tonometry (breast softness)
  * Baker Capsular Contracture grade
  * Aesthetic outcome (using Likert score) This will be assessed by the clinical researcher, and independently assessed using the medical photographs, with the assessor blinded to the reconstruction technique

Assessment of Contracture Using the Baker Breast Contracture Scale, the researcher will assess the Baker Grade for each breast to assess the level of capsular contracture.

Baker Grade Parameters I the breast is normally soft and looks natural II the breast is a little firm but looks normal III the breast is firm and looks abnormal IV the breast is hard, painful, and looks abnormal

Inclusion Criteria

* Patients age 18 years or older at the time of surgery.
* Patients who have undergone immediate Implant-based breast reconstruction with or without Strattice™ with a minimum follow-up of six months.
* Patients capable of providing informed consent.

Exclusion Criteria

* Patients who have had an immediate implant-based breast reconstruction with an alternative brand of matrix/mesh to Strattice™.
* Patients who have had a flap based-reconstruction with implant.
* Delayed reconstructions.

Study Size and Statistical Analysis

* From three large breast units across the UK, we shall aim to recruit a maximum of 400 patients to the prospective part of the study.
* Statistical Analysis will be performed in collaboration with Dr Julie Morris, Honorary Senior Lecturer, Department of Medical Statistics. SPSS 15 will be used to analyse the data.

Study Sites:

University Hospital of South Manchester Newcastle Upon Tyne Hospitals NHS Trust Bradford Teaching Hospitals NHS Foundation Trust

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older at the time of surgery.
* Patients who have undergone immediate Implant-based breast reconstruction with or without Strattice™ with a minimum follow-up of six months.
* Patients capable of providing informed consent.

Exclusion Criteria:

* Patients who have had an immediate implant-based breast reconstruction with an alternative brand of matrix/mesh to Strattice™.
* Patients who have had a flap based-reconstruction with implant.
* Delayed reconstructions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients age 18 years or older at the time of surgery.
  * Patients who have undergone immediate Implant-based breast reconstruction with or without Strattice™ with a minimum follow-up of six months.
  * Patients capable of providing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2016-08-19 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients planned loss of implant within 12 months of immediate reconstruction | 12 months

SECONDARY OUTCOMES:
Quality of Life questionnaire | 8 years
In-patient treatment costs | 8 years
Ipsilateral Revision rates | 1-8 years
Cosmesis | 1-8 years
  Cosmesis domains of Breast-Q quality of life questionnaire and likert 1-5 scale
Breast Reconstruction softness | 1-8 years
  Using tonometric measurement of breast softness
Regional pain | 1-8 years
  Using pain domain of Breast-Q Quality of Life questionnaire
loco-regional cancer recurrence | 1-8 years
Morbidity | 1-8 years

OTHER OUTCOMES:
Effect of Radiotherapy | 1-8 years
  Patients will be recorded as to whether they have or have not received radiotherapy. Effect of radiotherapy on the primary and secondary outcome measures will be compared between and within groups

CONTACTS AND LOCATIONS:
Overall Officials: Richard Johnson, Principal Investigator — University Hospital of South Manchester